CLINICAL TRIAL: NCT04675892
Title: Resection of One or Both Slips of the Flexor Digitorum Superficialis Tendon for Cases of Severe Trigger Fingers. a Randomized Prospective Single Center Study
Brief Title: Resection of Flexor Digitorum Superficialis Tendon for Severe Trigger Fingers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Thierry Christen, Principal investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-01270
Record Dates: First submitted 2020-11-20; First posted 2020-12-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-02

CONDITIONS: Trigger Finger; Stenosing Tenosynovitis
Keywords: trigger finger; stenosing flexor tenosynovitis
MeSH Terms: conditions — Trigger Finger Disorder; Tendon Entrapment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants were randomized in two groups according to a computer-generated list ranging from 01 to 60 (www.randomization.com). Surgery was then performed according to the method chosen by randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A1 pulley group (Active Comparator): A1 pulley division only
  Interventions: Procedure: A1 pulley division
- A1 pulley + FDS group (Experimental): Combination of A1 pulley division and excision of one or both slips of the flexor digitorum superficialis tendon
  Interventions: Procedure: A1 pulley division + Resection of one or both slips of the FDS tendon

INTERVENTIONS:
Procedure: A1 pulley division — Local anesthesia with 5-10 ml of solution required (90 % lidocaine 1 % with 1 ug epinephrine, 10 % sodium bicarbonate 8.4 %).
  Division of the A1 pulley.
  Wound closure with absorbable sutures and application of a light dressing.
  Arms: A1 pulley group
Procedure: A1 pulley division + Resection of one or both slips of the FDS tendon — Local anesthesia with 5-10 ml of solution required (90 % lidocaine 1 % with 1 ug epinephrine, 10 % sodium bicarbonate 8.4 %).
  Division of the A1 pulley.
  Palmar Bruner incision over the PIP joint. Distal dissection and resection of one or both slips of the FDS tendon.
  Wound closure with absorbable sutures and application of a light dressing.
  Arms: A1 pulley + FDS group

SUMMARY:
The purpose of this study is to compare the effectiveness of resection of one or both slips of the flexor digitorum superficialis tendon versus the A1 pulley division.

DETAILED DESCRIPTION:
The preoperative visit occurred a number of weeks or months prior to surgery. Surgeons from the Centre de la main at the CHUV in Lausanne recruited the subjects during their consultations. During this initial visit, the patient was asked about his problem, his general health and a clinical examination (including range of motion of finger joints, pulp-to-palm distance, pain evaluated with a VAS) was performed. Once the diagnosis of trigger finger was established, the inclusion and exclusion criteria were evaluated. If the eligibility criteria were fulfilled, the patients were offered to be part of the study. They received oral and written information about the study and the surgeons gave further explanation if needed.

On the surgery day, the signed consent form was recovered. Participants were randomized in two groups according to a computer-generated list ranging from 01 to 60 (www.randomization.com). Surgery was then performed according to the method chosen by randomization. The possible occurrence of adverse effects during surgery was monitored. All information was recorded on the case report forms.

The first postoperative visit occurred 1 week ± 3 days after surgery. The surgeons evaluated the wound to exclude the presence of postoperative complication (infection, hematoma, nerve or tendon injury) and answer any question the patient could have. Range of motion and pain were recorded. All information was recorded on the case report forms.

The second postoperative visit occurred 4 weeks ± 5 days after surgery. The appointment was conducted in the same way as the previous one.

Patients could choose to be withdrawn from the study at any point. The follow-up was similar to that of patients included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) with a flexor tendon tenosynovitis of a finger resulting in a decreased range of motion of the PIP joint (defined with a palm-to-pulp distance ≥0mm and/or flexion contracture ≥15°).

Exclusion Criteria:

* Minors (<18 years old).
* PIP joint contracture resulting from another illness than stenosing flexor tenosynovitis (for example: rheumatoid arthritis) or caused by a traumatic event.
* Contraindications to any surgery: presence of a severe coagulation disorder, immunosuppression or decompensated psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in total active finger motion in degrees | Preoperative (days to weeks prior to surgery), 4 weeks after surgery
  Change in preoperative and postoperative overall range of motion of the finger joints in degrees

SECONDARY OUTCOMES:
Change in with the visual analog scale | Preoperative (days to weeks prior to surgery), 4 weeks after surgery
  Change in pain with the visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No